CLINICAL TRIAL: NCT01723449
Title: Predictors for Admission to Emergency Department More Than 48 Hours
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Christian Backer Mogensen, assistant professor, University of Southern Denmark
Other Study IDs: SHS-ED-01-2012
Record Dates: First submitted 2012-10-24; First posted 2012-11-07 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Length of Admission

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In Demark acutely admitted patients are supposed to stay in the Emergency Department (ED) bed ward if the anticipated duration of stay is less than 48 hours.

However, it is not a trivial matter to estimate duration of stay for emergency patients. a number of factors affect this, eg. social background, disease, hospital organisation.

The aim of this study is to analyse whom are the best among the health staff to predict the length of stay: ED nurses, admitting doctors og the specialist, and to analyse if a number of variables can be used to improve the prediction.

ELIGIBILITY:
Inclusion Criteria:

all patients admitted to the Emergency Department -

Exclusion Criteria:

Children less than 15 years patients transferred from other hospitals

-

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all admissions to Emergency department
Sampling Method: Probability Sample
Enrollment: 730 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
length of admission in hours | admission to discharge
  participants will be followed for the duration of hospital stay, an expected average of 76 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Aabenraa Sygehus Emergency Department, Aabenraa, Denmark